CLINICAL TRIAL: NCT00353951
Title: Genomics to Combat Resistance Against Antibiotics in Community-Acquired LRTI in Europe: GRACE. Workpackage 8. An Observational Study of Cough / Lower Respiratory Tract Infection (LRTI) in Primary Care
Brief Title: An Observational Study of Cough / Lower Respiratory Tract Infection (LRTI) in Primary Care
Status: Completed | Type: Observational
Sponsor: Cardiff University (Other)
Collaborators: European Commission (Other); University of Southampton (Other); Universiteit Antwerpen (Other); Utrecht University (Other)
Other Study IDs: GRACE-01
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Cough; Lower Respiratory Tract Infection (LRTI); Chest Infection
Keywords: primary care; lower respiratory tract infection; antibiotics; cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The overall objective of GRACE is to combat the resistance of drugs that kill bacteria and other germs (antimicrobial) through integrating centres of research excellence and using the study of the entire DNA in a cell (genomics) to most appropriately investigate and manage community-acquired LRTI.

Grace-01 is the first study to be undertaken as part of GRACE and the aims of this study are to describe the presentation, diagnosis, investigation, management and outcomes for people with cough / chest infection in general medical practice in 13 primary care networks in 12 countries in Europe.

DETAILED DESCRIPTION:
GRACE is a Network of Excellence focusing on the complex and controversial field of community-acquired lower respiratory tract infections (LRTI), which is one of the leading reasons for seeking medical care. It is funded through Funding Program 6 of the European Union. The prescription of antibiotics for LRTI accounts for a major proportion of antibiotics used in the community, and contributes to the rising prevalence of resistance among major human pathogens. The overall objective of GRACE is to combat antimicrobial resistance through integrating centres of research excellence and exploiting genomics in the investigation and management of community-acquired LRTI

The first study undertaken as part of GRACE is GRACE-01, an observational study, which aims to describe the presentation, management (evaluation and treatment decisions) and outcomes for people with cough / chest infection in general medical practice in 13 primary care networks in Europe. This will be an observational study of current practice involving no experimental procedures or interventions.

Other objectives Of GRACE-01 are:

1. To describe variation in management of cough / chest infection including antibiotic prescribing in primary care between, and within, selected European countries in order to explain how good practice could be made explicit and generalised.
2. To identify priorities for intervention studies aimed at enhancing antibiotic prescribing for community acquired cough / chest infection and other aspects of management.
3. To contribute to developing interventions aimed at enhancing antibiotic prescribing and other aspects of management of community-acquired cough / chest infection that are applicable across the European Union (EU), and also to interventions that are relevant to unique local situations within Europe.

There will be two recruitment periods, one beginning on the second of October 2006 or soon thereafter and a second beginning on the first of February 2007 or soon thereafter. The goal is for each of the 13 participating European networks to recruit a total of 150 patients during each of these recruitment periods.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over.
* With acute or worsened cough with a duration of up to and including 28 days, or a clinical presentation that suggests a lower respiratory tract infection.
* Consulting for the first time within this illness episode.
* Seen within normal consulting hours.
* Able to fill out study materials.
* Who have provided written, informed consent to participate.

Exclusion Criteria:

* Previous study participants.
* Immunocompromised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3402 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Butler, FRCGP CCH MD, Principal Investigator — Cardiff University
Locations (1):
- GRACE Network in Cardiff, Cardiff, United Kingdom

REFERENCES:
- [Derived] Nuttall J, Hood K, Verheij TJ, Little P, Brugman C, Veen RE, Goossens H, Butler CC. Building an international network for a primary care research program: reflections on challenges and solutions in the set-up and delivery of a prospective observational study of acute cough in 13 European countries. BMC Fam Pract. 2011 Jul 27;12:78. doi: 10.1186/1471-2296-12-78. PMID 21794112
- [Derived] Butler CC, Kelly MJ, Hood K, Schaberg T, Melbye H, Serra-Prat M, Blasi F, Little P, Verheij T, Molstad S, Godycki-Cwirko M, Edwards P, Almirall J, Torres A, Rautakorpi UM, Nuttall J, Goossens H, Coenen S. Antibiotic prescribing for discoloured sputum in acute cough/lower respiratory tract infection. Eur Respir J. 2011 Jul;38(1):119-25. doi: 10.1183/09031936.00133910. Epub 2011 Mar 15. PMID 21406512
- [Derived] Stanton N, Hood K, Kelly MJ, Nuttall J, Gillespie D, Verheij T, Little P, Godycki-Cwirko M, Goossens H, Butler CC. Are smokers with acute cough in primary care prescribed antibiotics more often, and to what benefit? An observational study in 13 European countries. Eur Respir J. 2010 Apr;35(4):761-7. doi: 10.1183/09031936.00168409. Epub 2009 Dec 23. PMID 20032009
- [Derived] Butler CC, Hood K, Verheij T, Little P, Melbye H, Nuttall J, Kelly MJ, Molstad S, Godycki-Cwirko M, Almirall J, Torres A, Gillespie D, Rautakorpi U, Coenen S, Goossens H. Variation in antibiotic prescribing and its impact on recovery in patients with acute cough in primary care: prospective study in 13 countries. BMJ. 2009 Jun 23;338:b2242. doi: 10.1136/bmj.b2242. PMID 19549995